CLINICAL TRIAL: NCT00730977
Title: A Pilot Study to Investigate the Tolerability of Inhaled Dry Powder Mannitol (IDPM) Administered Via a Novel Dry Powder Inhaler Device in Healthy Individuals and Subjects With Bronchiectasis.
Brief Title: A Pilot Study to Investigate Administration of Mannitol Via a Novel Dry Powder Inhaler Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Brett Charlton, Pharmaxis Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DPM-DEV-101b
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Healthy; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): single arm, open label, 4 doses tested.
  Interventions: Drug: dry powder inhaled mannitol

INTERVENTIONS:
Drug: dry powder inhaled mannitol — single doses of 40 mg, 70 mg and 100 mg

SUMMARY:
A novel dry powder inhaler device will be used to administer mannitol to healthy subjects and subjects with bronchiectasis in single doses higher than previously given.The main objective is to assess tolerability of these doses using the new device.

ELIGIBILITY:
Inclusion Criteria:

* healthy or bronchiectatic; 18 years and over

Exclusion Criteria:

* uncontrolled asthma, unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
tolerability | immediately and 10 mins post dose

SECONDARY OUTCOMES:
respiratory symptoms, FEV1 | pre-dose, immediately and 10 mins post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Prince Alfred Hospital, Sydney, Australia